CLINICAL TRIAL: NCT00709228
Title: PREDICT - Prospective Observational Study Of A Cohort Of Naïve Patients With Chronic Hepatitis C Infected With Hepatitis C Virus Genotype 1 Low Viral Load (HCV LVL G1) And Treated With Peg-Intron 1.5 ug/Kg/Week Plus Rebetol 800-1200 mg/Day Who Achieved A Negative HCV-RNA At Week 4 and at Week 24
Brief Title: Study of Patients With Chronic Hepatitis C Infected With HCV LVL G1 and Effect of Peg-Intron Plus Rebetol Treatment (Study P04793)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04793
Record Dates: First submitted 2008-06-23; First posted 2008-07-03 (Estimated); Results first posted 2010-02-22 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for PCR
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PegIntron plus Rebetol: Those with chronic Hepatitis C infected with HCV LVL G1
  Interventions: Drug: PegIntron; Drug: Rebetol

INTERVENTIONS:
Drug: PegIntron — 1.5 ug/kg/week
  Other Names: SCH 054031
Drug: Rebetol — 800-1200 mg/day
  Other Names: SCH 18908

SUMMARY:
To determine the relapse rate at 24 weeks follow up in Hepatitis C Virus Genotype 1 Low Viral Load (HCV LVL G1) patients treated for 24 weeks with Peg Intron and Rebetol who are Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) negative at treatment week 4 and week 24. To determine the proportion of patients (%) with sustained virological response at 24 weeks post follow up treatment.

DETAILED DESCRIPTION:
Approximately 500 patients from about 100 sites to be identified as HCV LVL G1 patients

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* 18 years or older, either gender, any race
* Must have Hepatitic C Virus Low Viral Load [LCV LVL] (positive, but <600,000 IU/mL on the assay used by the individual study site. Only Hepatitis C Virus-Ribonucleic acid/quantitative polymerase chain reaction [HCV-RNA/qPCR] assays with results in IU/ml are acceptable) AND been diagnosed with Genotype 1
* Subject considered suitable for treatment per local label
* Investigator considers suitable and subject consents to be treated

Exclusion Criteria:

* Does not show negative polymerase chain reaction [PCR] at week 4
* Pregnant women or those who plan to become pregnant or sexual partners of women who plan to become pregnant
* Subject does not qualify based on contra-indication, special warning, special population, and/or pregnancy & lactation section of the Summary of Product Characteristics [SmPC]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

REFERENCES:
- [Result] Craxi A, Koutsounas S, Ogurtsov P, Chemello L, Maticic M, Torras J, Diago M, Tartaglione MT, Witthoeft T, Yu X, Faruqi R, Chaudhri E, Pedicone LD, Zuckerman E. Peginterferon alfa-2b plus weight-based ribavirin for 24 weeks in patients with chronic hepatitis C virus genotype 1 with low viral load who achieve rapid viral response. J Viral Hepat. 2012 Feb;19(2):e120-5. doi: 10.1111/j.1365-2893.2011.01515.x. Epub 2011 Sep 19. PMID 22239509

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIntron Plus Rebetol: Those with chronic Hepatitis C infected with Hepatitis C Virus Genotype 1 Low Viral Load (HCV LVL G1) and treated withPeg-Intron 1.5 μg/kg/week plus Rebetol (ribavirin) 800-1200 mg/day who achieved a negative Hepatitis C Virus-Ribonucleic Acid (HCV-RNA) at Week 4 and at Week 24
Period: Overall Study
Arm/Group | PegIntron Plus Rebetol
Started | 496
Completed | 164 (Number completed is defined as participants who completed the follow-up period.)
Not Completed | 332
Not completed — Not treated | 14
Not completed — Eligibility criteria not met | 281
Not completed — Adverse events | 2
Not completed — Discontinued treatment | 14
Not completed — Did not enter follow-up | 4
Not completed — Discontinued follow-up | 5
Not completed — Disease progression | 1
Not completed — Lost to Follow-up | 6
Not completed — Non-compliance | 5

BASELINE CHARACTERISTICS:
Groups:
- PegIntron Plus Rebetol: Those with chronic Hepatitis C infected with Hepatitis C Virus Genotype 1 Low Viral Load (HCV LVL G1) and treated withPeg-Intron 1.5 μg/kg/week plus Rebetol (ribavirin) 800-1200 mg/day who achieved a negative HCV-RNA at Week 4 and at Week 24 (n = 170)
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of HCV LVL G1 Participants Who Relapsed
Description: Relapse was defined as undetectable Hepatitis C virus-ribonucleic acid (HCV-RNA) at End of Treatment, but detectable HCV-RNA at Follow-up Week 24.
Time Frame: Week 24 of follow-up
Population: The 165 participants analyzed is from the efficacy evaluable population (170) minus 5 subjects who did not have follow-up data.
Measure: Number; unit: Participants
Arm/Group | PegIntron Plus Rebetol
Number analyzed (Participants) | 165
Participants | 16
Statistical Analysis 1: Comparison: PegIntron Plus Rebetol; Test type: Superiority or Other; simple proportion = 0.097, 95% CI 2-sided [0.06 to 0.15]

ADVERSE EVENTS:
Description: Number analyzed is the number of treated participants (482 of the 496 screened).
Arm/Group | PegInton Plus Rebetol
Serious Adverse Events (participants affected / at risk) | 11/482
Other Adverse Events (participants affected / at risk) | 0/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegInton Plus Rebetol (N=482)
PERICARDITIS (Cardiac disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
ABSCESS NECK (Infections and infestations) | 1 (1)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1)
AGGRESSION (Psychiatric disorders) | 1 (1)
PERSONALITY DISORDER (Psychiatric disorders) | 1 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Lead investigator agrees not to publish or publicly present any interim results of the Study without prior written consent of the sponsor. Lead investigator further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication, which report any results of the Study. Sponsor shall have the right to review and comment on any presentation, including editorial rights.